# Study Protocol and Statistical Analysis Plan — Cover Page

#### **Official Study Title:**

Assessing the Utility of a Remote Patient Monitoring Platform for Improving CPAP Adherence for Obstructive Sleep Apnea

## **NCT Number:**

To be assigned

#### **Date of Document:**

February 5, 2024

## Sponsor:

MonitAir LLC

#### **Collaborator:**

BetterNight

#### **Principal Investigators:**

- Dominic Munafo, MD
- Edward Mezerhane, MD

### **Study Location:**

BetterNight clinical network (United States)